CLINICAL TRIAL: NCT05000645
Title: Grocery Delivery and Healthy Weight Gain Among Low-income Pregnant Young Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Tammy Chang, Assistant Professor of Family Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00190614; 1R01HD101522 (NIH)
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; Weight Gain
Keywords: WIC; Low-income; Diet; Sugar sweetened beverages; Grocery delivery
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Women, Infants, and Children (WIC) (No Intervention): Usual WIC counseling and food benefits for use in person at approved grocery stores.
- WIC + grocery delivery (Experimental): Usual WIC counseling and food benefits, as well as twice-monthly home deliveries of WIC-approved foods.
  Interventions: Behavioral: Grocery delivery
- WIC + grocery delivery + unsweetened beverage delivery (Experimental): Usual WIC counseling and food benefits as well as twice-monthly home deliveries of WIC-approved foods PLUS unsweetened beverages to replace their current sugar-sweetened beverages (SSB) intake.
  Interventions: Behavioral: Grocery delivery; Behavioral: Unsweetened beverage delivery

INTERVENTIONS:
Behavioral: Grocery delivery — Each food delivery will contain approximately $35 worth of fresh fruits, vegetables, dairy products, and whole grain foods. These foods are not meant to supplant regular meals, rather make healthy eating more convenient.
  Arms: WIC + grocery delivery; WIC + grocery delivery + unsweetened beverage delivery
Behavioral: Unsweetened beverage delivery — Participants will receive unsweetened beverages to replace normal sugar-sweetened beverage intake.
  Arms: WIC + grocery delivery + unsweetened beverage delivery

SUMMARY:
This project will increase knowledge about how a simple intervention, grocery delivery, impacts weight gain and diet among low-income pregnant young women. Results can then be used to support other pregnant young women.

DETAILED DESCRIPTION:
The overall aim of this study is to determine whether an intervention that facilitates receipt of healthy food and unsweetened beverages will promote healthy weight gain and improve diet quality among pregnant young women age 14-26 living in Michigan. This hypothesis will be tested in a three-arm randomized controlled trial (RCT) using a parallel design; Arm 1: Usual WIC (Control), Arm 2: Usual WIC + Delivery of WIC-approved food, Arm 3: Usual WIC + Delivery of WIC-approved food PLUS unsweetened beverages. Three arms are necessary because our goal is to make three distinct comparisons. First, we need to determine the effect of food delivery (Arm 2) compared to usual WIC (Arm 1). Second, we need to determine the combined effect of food plus unsweetened beverage delivery (Arm 3) compared to usual WIC (Arm 1). Finally, we need to evaluate the effect of food delivery (Arm 2) compared with food plus unsweetened beverage delivery (Arm 3) to determine the individual impact of replacing SSBs, a major contributor to excessive pregnancy weight gain in our population. Our study does not assess the impact of delivering only unsweetened beverages compared to usual WIC because the potential policy implication is the delivery of WIC benefits. A widespread program that only delivers unsweetened beverages is not likely.

Upon completion of baseline screening and assessments, 570 pregnant young women will be randomly assigned to either the control group or one of the two experimental groups. Enrollment in the study is rolling and starts as early as possible in the pregnancy (must be before 21 weeks gestation). The intervention period begins at enrollment and continues to the end of pregnancy/birth. Thus, each participant will be enrolled for approximately seven months post-randomization. During the intervention period, all groups will receive usual WIC food, nutritional assessment, and counseling benefits, including monthly intensive nutritional counseling sessions based on a state-approved curriculum with trained nutritionists and peer counselors.

* The control group (Arm 1) will receive usual WIC counseling and food benefits loaded onto their electronic benefits card (EBT) for them to use in person at approved grocery stores.
* The first experimental group (Arm 2) will receive usual WIC counseling and food benefits, as well as twice-monthly home deliveries of WIC-approved foods.
* The second experimental group (Arm 3) will receive usual WIC counseling and food benefits as well as twice-monthly home deliveries of WIC-approved foods PLUS unsweetened beverages to replace their current SSB intake.

The primary outcome is weight gain during pregnancy as defined by the Institute of Medicine (IOM)/National Academy of Medicine (NAM) Guidelines. Secondary outcomes include Healthy Eating Index (HEI) scores and dietary intake of fruits, vegetables, whole grains, and SSBs; infant birth weight; and prenatal and delivery complications identified through postpartum medical record review (e.g., small/large for gestational age, gestational diabetes, hypertensive disorders, operative delivery).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤ 20 weeks
* Text message capability
* Healthy singleton pregnancy
* Nulliparous
* Consume sugar sweetened beverages (SSBs)
* Living within delivery zone of a grocery delivery service

Exclusion Criteria:

* Non-English speaking
* Participants who live at the same address
* Physical, mental, or cognitive handicaps that prevent participation
* High risk pregnancy requiring specialized care (including pre-existing diabetes)

Ages: 14 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 570 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Weekly weight gain in pregnancy | Up to delivery, approximately 40 weeks
  Frequency of weight categorizations, categorized as above, below, or within Institute of Medicine/National Academy of Medicine (IOM/NAM) guidelines, will be assessed. Data collected from BodyTrace scale and calculated as weight for a particular week minus pre-pregnancy weight.
Total weight gain in pregnancy | At delivery, approximately 40 weeks
  Frequency of weight categorizations, categorized as above, below, or within Institute of Medicine/National Academy of Medicine (IOM/NAM) guidelines will be assessed. Data collected from BodyTrace scale and calculated as end of pregnancy weight minus pre-pregnancy weight.

SECONDARY OUTCOMES:
Dietary Quality as measured by the Healthy Eating Index (HEI) Score | Up to delivery, approximately 40 weeks
  Dietary recall data collected via the ASA24 (Automated Self-Administered 24-Hour) Dietary Recall Survey will be used to determine continuous HEI scores. ASA24 data are collected twice at enrollment, twice in second trimester, and twice in third trimester and used in pairs to calculate 3 HEI scores per participant. The HEI uses a scoring system to evaluate a set of foods. The scores range from 0 to 100 with higher scores correlating to higher diet quality.
Occurrence of prenatal complications | Delivery, approximately 40 weeks
  Frequency of prenatal complications will be assessed. Complications are collected from mother's medical record examples include gestational diabetes and hypertensive disorders.
Occurrence of delivery complications | Delivery, approximately 40 weeks
  Frequency of delivery complications will be assessed. Complications are collected from mother's medical record and include operative delivery, shoulder dystocia, and postpartum hemorrhage.
Baby birth weight | Delivery, approximately 40 weeks
  Collected from mother's medical record and will be categorized as small, appropriate, or large for gestational age based on weight percentiles (small < 10th percentile, appropriate ≥ 10th percentile and ≤ 90th percentile, large > 90th percentile).

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Chang, MD, MPH, MS, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waselewski M, Plegue M, Sonneville K, Resnicow K, Ghumman A, Ebbeling C, Mahmoudi E, Sen A, Wolfson JA, Chang T. Grocery Delivery to Support Healthy Weight Gain Among Pregnant Young Women With Low Income: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Aug 5;11(8):e40568. doi: 10.2196/40568. PMID 35930351